CLINICAL TRIAL: NCT04856852
Title: Iodine-125 Brachytherapy Together With Chemotherapy Compared With Surgical Resection Followed by Concomitant Radiochemotherapy in Patients With Newly Diagnosed Glioblastoma，a Randomized, Open-label, Multi-center Clinical Trial
Brief Title: Iodine-125 Brachytherapy Together With Chemotherapy in Patients With Newly Diagnosed Glioblastoma
Acronym: IBCNG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC-SRC-20201119; 2019YFE0120100 (Other Grant/Funding Number: MOST)
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Iodine-125; Surgical resection; Radiochemotherapy; Chemotherapy; Radiation
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iodine-125+Chemotherapy (Experimental): Iodine-125; Temozolomide
  Interventions: Other: Iodine-125+Chemotherapy
- Surgical resection+Radiochemotherapy (Active Comparator): Surgical resection; Radiotherapy; Temozolomide:
  Interventions: Other: Surgical resection+Radiochemotherapy

INTERVENTIONS:
Other: Iodine-125+Chemotherapy — Iodine-125: Iodine-125 if necessary, 0.6-0.8mCi, PD:120-150Gy Temozolomide: 75 mg per square meter of body-surface area per day, 7 days per week,42 days.
  Other Names: Iodine-125+Temozolomide
  Arms: Iodine-125+Chemotherapy
Other: Surgical resection+Radiochemotherapy — Surgical resection: Maximal surgical resection, including gross total resection, subtotal resection, and partial resection.
  Radiation: total 60 Gy, 2 Gy per daily fraction (Monday to Friday) for 6 weeks. Temozolomide: 75 mg per square meter of body-surface area per day, 7 days per week,42 days.
  Other Names: Surgical resection+Radiotherapy+Temozolomide
  Arms: Surgical resection+Radiochemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Iodine-125 brachytherapy together with chemotherapy compared with surgical resection followed by concomitant radiochemotherapy in patients with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
This is a prospective, multicentric open-label trial to evaluate the efficacy and safety of Iodine-125 brachytherapy together with chemotherapy compared with surgical resection followed by concomitant radiochemotherapy in patients with newly diagnosed glioblastoma.

The primary efficacy outcome was evaluated with progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of glioblastoma confirmed by histology
* 2. Age: 18-75 years old
* 3. Single lesion located in one hemisphere with a diameter between 2 and 6 centimeters
* 4. No prior anticancer therapy for glioblastoma besides biopsy.
* 5. ECOG PS：0-2 point

Exclusion Criteria:

* 1. Infra-tentorial tumor or tumor involves the ependymal surface.
* 2. Nonmeasurable disease.
* 3. Evidence of uncontrolled intracranial pressure.
* 4. Severe heart, brain, and lung diseases.
* 5.Severe hepatic or renal dysfunction.
* 6. Uncontrolled, active infection.
* 7. Severe clotting dysfunction.
* 8. Pregnant.
* 9. Uncontrolled hypertension.
* 10. Participated in any other clinical treatment trial within 4 weeks before randomization.
* 11. Severe vascular diseases within 6 months before randomization.
* 12. Participants who received major surgical treatment within 4 weeks or were expected to be treated during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-06-28 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2.5 years after randomization
  PFS is defined as the time from randomization to progression or death from any causes. Progression is defined as the RANO Criteria indicated.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2.5 years after randomization
  OS is defined as the time from randomization to death from any causes.
Survival rates at 6 months and 1 year | at 6 months and 1 year after operation respectively
  The survival rates were measured at 6 months and 1 year
EORTC QLQ-C30 | 2.5 year after randomization
  The Quality of life is measured with EORTC QLQ-C30 (The European Organization for Research and Treatment of Cancer Core Quality of Life questionnaire). The EORTC QLQ-C30 is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items.
ECOG Performance Status | 2.5 year after randomization
  ECOG PS (Eastern Cooperative Oncology Group, performance status) is to assess how a patient's disease is progressing, and how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. The scale is from 0 to 5. Higher scores mean a worse outcome.
Complications | within 1 week after operation
  Complications 1 week after operation were assessed. The complications after operation include headache, nausea, vomit, myodynamia, seizer, and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaokun Hu, MD, Principal Investigator — The Affiliated Hospital of Qingdao University

IPD SHARING:
Plan to Share IPD: No